CLINICAL TRIAL: NCT02642575
Title: Automated Folliculometry Using Five-Dimensional Ultrasound
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rehab Mohamed Abdelrahman, Principal Investigator, Ain Shams University
Other Study IDs: 5D Folliculometry
Record Dates: First submitted 2015-12-28; First posted 2015-12-30 (Estimated); Results first posted 2017-05-08 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-05

CONDITIONS: Automated Folliculometry Using Five-Dimensional Ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of the study to evaluate Five-Dimensional Ultrasound in automated measurement of ovarian follicles with controlled ovarian stimulation in contrast to the conventional 2D ultrasound

DETAILED DESCRIPTION:
This is a Prospective pilot study that will be performed at the Fetal Care Unit at Ain Shams University Maternity Hospital.

72 women will be recruited from the the Fetal Care Unit who will fulfill the inclusion criteria. They will be counseled to be included into the study.

All cases will be subjected to:

full history taking including patient's age, parity,last menstrual period , past history of medical disorders, clinical examinations (General and abdominal).

Two-Dimensional Ultrasound and Five-Dimensional Ultrasound will be done for all cases for assessment of ovarian follicles after controlled ovarian stimulation by clomid 50 mg5×2×1 The automated software allows for automated three-dimensional follicular measurement.The software then analyzes the volume and automatically identifies all of the follicles in the ovary. The software also automatically generates several volumetric parameters of each and every identified follicle.

ELIGIBILITY:
Inclusion Criteria:

* all women between 25 to 35 years of age
* all women have a normal body mass index(18-25kg/M^2)
* regular menstrual cycles
* all women would be receiving ovarian stimulation using clomiphene citrate (clomid 50 mg) for ≥5 days starting from 5th day of the cycle then they will be scanned by the same physician using Two Dimensional Ultrasound then Five Dimensional Ultrasound U/S

Exclusion Criteria:

1. medical disorders
2. obesity. BMI>30

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This is a Prospective pilot study that will be performed at the Fetal Care Unit at Ain Shams University Maternity Hospital.
  67 women will be recruited from the the Fetal Care Unit who will fulfill the inclusion criteria. They will be counseled to be included into the study.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2015-12; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
The aim of the study to evaluate Five-Dimensional Ultrasound in automated measurement of ovarian follicles with controlled ovarian stimulation in contrast to the conventional 2D ultrasound

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Prospective pilot study that was performed at the Fetal Care Unit at Ain Shams University Maternity Hospital from January 2016 to august 2016.
  67 women were recruited from the Fetal Care Unit who fulfilled the inclusion criteria. Verbal consent was obtained from participants who were included into the study.
Groups:
- Folliculometry in Women With Unexplained Infertility: 67 women who were recruited from the Fetal Care Unit who fulfilled the inclusion criteria, would be receiving ovarian stimulation using clomiphene citrate (clomid 50 mg) for ≥5 days starting from 5th day of the cycle then they will be scanned by the same physician using Two Dimensional Ultrasound then Five Dimensional Ultrasound.
Period: Overall Study
Arm/Group | Folliculometry in Women With Unexplained Infertility
Started | 67
Completed | 67
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 67 women were recruited from the Fetal Care Unit who fulfilled the inclusion criteria. Verbal consent was obtained from participants who were included into the study.
Arm/Group | Folliculometry in Women With Unexplained Infertility
Number analyzed (Participants) | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 67
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67
  Male | 0
Region of Enrollment [Number; unit: Count of Participants]
  Egypt | 67

OUTCOME MEASURES:

1. Primary Outcome: The Mean Follicular Diameter by Two-Dimensional Ultrasound
Description: All women would be receiving ovarian stimulation using clomiphene citrate (clomid 50 mg) once daily for 5 days starting from 2nd day of the cycle then they will be scanned at 10th day by the same physician using Two Dimensional Ultrasound was done.
  Each follicle was assessed by measuring the maximal diameters on three orthogonal planes.
  The mean of three diameters was calculated.
Time Frame: 10th day of the menstrual cycle
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Folliculometry in Women With Unexplained Infertility
Number analyzed (Participants) | 67
mm | 8.41 (3.79)

2. Secondary Outcome: The Mean Follicular Diameter by Five-Dimensional Ultrasound
Description: All women would be receiving ovarian stimulation using clomiphene citrate (clomid 50 mg) once daily for 5 days starting from 2nd day of the cycle then they will be scanned at 10th day by the same physician using Five Dimensional Ultrasound was done.
  Five Dimensional Ultrasound automatically identifies hypoechogenic follicles within the captured ovarian volume and generates a set of measurements for each follicle. These measurements include the largest diameters in three orthogonal planes, the mean follicular diameter (MFD)
Time Frame: 10th day of the menstrual cycle
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Folliculometry in Women With Unexplained Infertility
Number analyzed (Participants) | 67
mm | 8.46 (3.89)

3. Secondary Outcome: The Volume-based Diameter (dV) of the Follicle by Five-Dimensional Ultrasound
Description: All women would be receiving ovarian stimulation using clomiphene citrate (clomid 50 mg) once daily for 5 days starting from 2nd day of the cycle then they will be scanned at 10th day by the same physician using Five Dimensional Ultrasound was done.
  Five Dimensional Ultrasound automatically identifies hypoechogenic follicles within the captured ovarian volume and generates a set of measurements for each follicle including the volume-based diameter (dV) of the follicle.
  The volume calculation is based on the voxel count within the identified follicle. It therefore represents a true measure of follicular volume.
Time Frame: 10th day of the menstrual cycle
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Folliculometry in Women With Unexplained Infertility
Number analyzed (Participants) | 67
mm^3 | 1193.29 (987.46)

ADVERSE EVENTS:
Time Frame: 1 year march 2016 to march 2017
Description: Two-Dimensional Ultrasound and Five-Dimensional Ultrasound were performed and adverse Events Adverse Events were assessed.
Arm/Group | Folliculometry in Women With Unexplained Infertility
Serious Adverse Events (participants affected / at risk) | 0/67
Other Adverse Events (participants affected / at risk) | 0/67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No